CLINICAL TRIAL: NCT01140035
Title: Intensive Insulin Therapy in Deceased Donors - to Improve Renal Allograft Function and Transplanted Allograft Outcomes
Brief Title: Intensive Insulin Therapy in Deceased Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California Transplant Donor Network (Network)
Responsible Party: Principal Investigator, Claus Niemann, Associate Professor of Anesthesia & Surgery, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R380T10586; HRSA R380T10586; HRSA (Other Grant/Funding Number: HRSA R380T10586)
Record Dates: First submitted 2009-09-10; First posted 2010-06-09 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Kidney Transplant
Keywords: Insulin; Deceased donors; Renal Allograft Function; Transplanted Allograft Outcomes
MeSH Terms: conditions — Insulin Resistance | interventions — Glycemic Control

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intensive insulin therapy (Experimental): Intensive insulin therapy with goal of glucose < 150 mg/dl
  Control group with standard insulin therapy with goal of glucose 180 mg/dl
  Interventions: Other: Administration of continuous insulin infusion for glycemic control in brain dead donors

INTERVENTIONS:
Other: Administration of continuous insulin infusion for glycemic control in brain dead donors — As per protocol
  Other Names: hyperglycemia

SUMMARY:
Every year in the US, there is a shortage of many thousands of kidneys needed for transplant. Furthermore, kidneys that are available and are transplanted often exhibit delayed or slow graft function (DGF and SGF, respectively), which lowers quality of life for patients and their families and requires significant additional medical care. These needs result in significant but preventable human suffering and health care spending. To address these needs, the investigators' project will test the use of intensive insulin therapy (IIT) in donors after neurological determination of death (DNDDs) as an intervention that will decrease acute kidney injury and improve renal function at the time of organ recovery. This should translate into a decreased incidence of DGF and SFG in recipients receiving organs from the IIT group. The investigators also expect to find a trend toward an increase in the number of organs available for transplant due to better organ protection in the DNDD. Taken together, these data can provide the requisite justification for a larger study that can be powered to evaluate the effect of IIT on increasing the number of kidneys available for transplantation.

There is evidence that brain death often leads to hyperglycemia that may negatively impacts the organs of DNDDs. These observations led us to conduct a retrospective study, in which the investigators found that hyperglycemia in DNDDs is indeed associated with decreased terminal renal function. Because it has been reported that intensive insulin therapy (ITT) is renoprotective in the ICU more than conventional insulin therapy (CIT), the investigators propose to evaluate the use of IIT on DNDDs to: (1) improve organ function, (2) reduce DGF in recipients, and (3) possibly increase the number of kidney available for transplant.

Methods: This is a prospective observational study to document the impact of IIT on acute kidney injury in DNDDS and on allograft function in recipients. DNDDs will be divided into two groups: CIT and IIT. In the first study, the investigators will evaluate the effect of ITT on biochemical parameters in blood samples that predict kidney health and function in DNDDs. All methods used in this proposal are well documented in the literature and established in the applicant's laboratory. In the investigators' second study, they will compare the effects of ITT in DNDDs on graft function in allograft recipients in terms of number of patients showing either DGF or SGF. Additionally, there is currently no established set of advanced biochemical criteria in DNDDs for predicting kidney function in recipients. The investigators will correlate the evaluated biochemical markers of kidney function and health in order to possibly develop more refined methods of predicting transplant success. Such a set of criteria would be useful for designing studies to systematically test additional interventions in DNDDs to further improve organ function before recovery and further increase the number of available organs.

Taken together, the results of this study may lead to new therapies that significantly improve patient outcomes while significantly reducing disease associated costs. These results can also set the stage for a follow on study for increasing the number of kidneys available for transplant.

ELIGIBILITY:
Inclusion Criteria:

* Deceased Organ Donors

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Renal Function in donor at the time of Aortic cross clamping | Between declaration of brain death and organ recovery (in average this period is 48 hrs)
  once organ donors are declared brain death and donor is consented for research, donor is randomized to control or experimental arm of study. The donation process between declaration of brain death and organ recovery is approximately 48 in our region.

SECONDARY OUTCOMES:
Graft function in kidney transplant recipient | Transplant surgery to 3 months post transplant
  Grafts of donors enrolled in the study will be followed in the recipient for 3 months. This time is sufficient to capture initial delayed graft function and short term renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Claus U Niemann, MD, Principal Investigator — UC San Francisco
Locations (1):
- U C San Francisco, San Francisco, California, United States